CLINICAL TRIAL: NCT00002779
Title: PHASE II TRIAL OF FLUDARABINE AND SANDOSTATIN FOR RELAPSED LOW-GRADE NON-HODGKIN'S LYMPHOMA
Brief Title: Fludarabine Plus Octreotide in Treating Patients With Relapsed Low-Grade Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-947851; NCCTG-947851; CDR0000064787 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 1999-11-01; First posted 2004-07-29 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Lymphoma
Keywords: Waldenström macroglobulinemia; recurrent small lymphocytic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma
MeSH Terms: conditions — Lymphoma; Waldenstrom Macroglobulinemia; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone | interventions — fludarabine phosphate; Octreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- fludarabine + octreotide (Experimental): Patients receive fludarabine IV over 10-30 minutes on days 1-5. Patients not currently receiving octreotide, receive a test dose of octreotide subcutaneously on day 1 during course 1 only and then receive octreotide intramuscularly monthly on day 1. Treatment repeats every 28 days for 4-6 courses. Patients then receive octreotide alone for 6-8 courses. Some patients may then receive another 12 courses of octreotide alone, for a total of 2 years of treatment. Patients are followed every 3 months for 5 years or until disease progression.
  Interventions: Drug: fludarabine phosphate; Drug: octreotide acetate

INTERVENTIONS:
Drug: fludarabine phosphate
Drug: octreotide acetate

SUMMARY:
RATIONALE: Drugs used in chemotherapy and hormone therapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of fludarabine plus octreotide in treating patients who have relapsed low-grade non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate and duration of response to fludarabine combined with octreotide and to octreotide alone in patients with relapsed indolent non-Hodgkin's lymphoma. II. Determine serum insulin-like growth factor-1 (IGF-1) and IGF-1 binding protein levels before and after treatment in this patient population. III. Determine somatostatin receptor subtypes in lymphoma biopsy samples from selected patients.

OUTLINE: Patients receive fludarabine IV over 10-30 minutes on days 1-5. Patients not currently receiving octreotide, receive a test dose of octreotide subcutaneously on day 1 during course 1 only and then receive octreotide intramuscularly monthly on day 1. Treatment repeats every 28 days for 4-6 courses. Patients then receive octreotide alone for 6-8 courses. Some patients may then receive another 12 courses of octreotide alone, for a total of 2 years of treatment. Patients are followed every 3 months for 5 years or until disease progression.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically diagnosed indolent non-Hodgkin's lymphoma (NHL) of 1 of the following types: Diffuse small lymphocytic cell Follicular small cleaved cell Follicular mixed small and large cleaved cell Mantle cell lymphoma/leukemia (intermediate differentiated lymphoma) Preferentially treated on protocol NCCTG-958053 when available Monocytoid B-cell Mucosa-associated lymphoid tissue (MALT) Lymphoplasmacytic lymphoma (Waldenstrom's macroglobulinemia) Histology documented by lymph node (or other mass) or bone marrow biopsy within 6 months prior to entry Relapsed after cytotoxic chemotherapy regimens At least 1 measurable lesion by palpation, chest x-ray, CT, or MRI, e.g.: Lymph node at least 1.5 x 1.5 cm by palpation Spleen at least 3 cm below left costal margin The following exclude: CNS involvement by positive CSF cytology or CT/MRI B- or T-cell chronic lymphocytic leukemia Hairy cell leukemia Mycosis fungoides Aggressive lymphoma

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Total bilirubin no greater than 2 times normal OR Direct bilirubin no greater than 1.0 mg/dL above normal Renal: Creatinine no greater than 2.0 times normal Cardiovascular: No uncontrolled congestive heart failure No uncontrolled hypertension No uncontrolled angina pectoris Other: No uncontrolled or active infection No AIDS or HIV antibody No second malignancy within 5 years except: Carcinoma in situ of the cervix Resected nonmelanomatous skin cancer Prostate cancer in remission following radical retropubic prostatectomy or radiotherapy Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Recovered from toxic effects of prior therapy Biologic therapy: See Disease Characteristics No concurrent interferon Chemotherapy: See Disease Characteristics No prior purine nucleoside analogues (e.g., fludarabine, pentostatin, or 2- chlorodeoxyadenosine) At least 3 weeks since prior chemotherapy (6 weeks since nitrosoureas) No other concurrent cytotoxic chemotherapy Endocrine therapy: No prior octreotide for lymphoma No concurrent corticosteriods except for Addison's disease Radiotherapy: Not specified Surgery: Not specified Other: No other concurrent investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 1998-02; Primary Completion 2000-07 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
response rate | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E. Witzig, MD, Study Chair — Mayo Clinic
Locations (20):
- United States (19):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Ochsner, New Orleans, Louisiana
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Quain & Ramstad Clinic, P.C., Bismarck, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Altru Health Systems, Grand Forks, North Dakota
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - CCOP - Geisinger Clinical and Medical Center, Danville, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
- Saskatchewan Cancer Agency, Regina, Saskatchewan, Canada